CLINICAL TRIAL: NCT04800224
Title: The Use of the Standardized Brazilian Green Propolis Extract (EPP-AF) as an Adjunct Treatment for Hospitalized COVID-19 Patients: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Brazilian Green Propolis Extract (EPP-AF) as an Adjunct Treatment for Hospitalized COVID-19 Patients (BeeCovid2)
Acronym: BeeCovid2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Apis Flora Industrial e Comercial Ltda (Unknown)
Responsible Party: Principal Investigator, Marcelo Augusto Duarte Silveira, MD, PhD, Principal Investigator, D'Or Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31099320.6.0000.0049
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Inflammation
Keywords: Propolis; Covid19; Anti-Inflammatory Agents; Immunoregulation
MeSH Terms: conditions — COVID-19; Inflammation | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The capsules will be coated, in opaque and equal packaging, so that the researchers involved in the care of patients could not distinguish between propolis and placebo. Neither the participants, nor the principal investigator, nor the health professionals involved in the care will know which group the patients will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients in the Placebo group will receive an identical number of capsules containing 900 mg / day of placebo (3 capsules of 100 mg each, divided into 3 daily doses); for 10 days.
  Interventions: Drug: Placebo
- Propolis (Active Comparator): Participants in the Propolis group will receive propolis EPP-AF at a dose of 900 mg / day (3 capsules of 100 mg each, divided into 3 daily doses); for 10 days.
  Interventions: Drug: Standardized Brazilian Green Propolis Extract

INTERVENTIONS:
Drug: Standardized Brazilian Green Propolis Extract — 900mg/day of Standardized Brazilian Green Propolis Extract for 10 days.
  Other Names: Propolis
  Arms: Propolis
Drug: Placebo — 900mg/day of Placebo for 10 days.
  Arms: Placebo

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) promotes challenging immune and inflammatory phenomena. Though various therapeutic possibilities have been tested against coronavirus disease 2019 (COVID-19), the most adequate treatment has not yet been established. Among candidate adjunct treatment options, propolis, produced by honey bees from bioactive plant exudates, has shown potential against viral targets and has demonstrated immunoregulatory properties.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of oral propolis as an adjunct treatment for SARS-CoV-2 infection, we designed a randomized, double-blind, placebo-controlled trial (Bee-Covid2) (The Use of Brazilian Green Propolis Extract (EPP-AF®) in Patients Affected by COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years;
* Diagnosis of coronavirus infection confirmed by polymerase chain reaction - reverse transcriptase testing;
* Symptoms started within 14 days of the randomization date

Exclusion Criteria:

* Pregnant or lactating women;
* Known hypersensitivity to propolis;
* Propolis use less than 30 days from the randomization date;
* Active cancer;
* Human immunodeficiency virus carriers;
* Patients undergoing transplantation of solid organs or bone marrow or who were using immunosuppressive medications;
* Bacterial infection at randomization, sepsis or septic shock related to bacterial infection at randomization;
* Impossibility of using the medication orally or by nasoenteral tube;
* Known hepatic failure or advanced heart failure (New York Heart Association [NYHA] class III or IV).
* End Stage Renal Disease (ESRD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 1-28 days
  Hospitalization time after randomization (in days)

SECONDARY OUTCOMES:
Percentage of participants with adverse events during the use of propolis or placebo | 1-28 days
  We will evaluate the presence or absence of symptoms related to the use of propolis or placebo.
Rate and severity of acute kidney injury during the study | 1-28 days
  Assess the degree of acute kidney injury according to KDIGO.
Renal replacement therapy. | 1-28 days
  Assess need or not for renal replacement therapy
Rate of need for vasopressor use. | 1-28 days
  Describe the time needed for vasopressors in days after randomization.
Intensive care unit (ICU) readmission | 1-28 days
  Rate of readmission to the ICU after randomization
Invasive oxygenation time | 1-28 days
  Assess the need for mechanical ventilation in days after randomization.
Need for Intra-Aortic Balloon Pump | 1-28 days
  Assess the need for Intra-Aortic Balloon Pump in days after randomization.
Need for Extracorporeal Oxygenation Membrane (ECMO) | 1-28 days
  Assess the need for Extracorporeal Oxygenation Membrane in days after randomization.

OTHER OUTCOMES:
Death | 1-28 days
  Assess mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Silveira, MD, PhD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- Hospital Sao Rafael, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are available on request from the corresponding author.

REFERENCES:
- [Background] Silveira MAD, Capcha JMC, Sanches TR, de Sousa Moreira R, Garnica MS, Shimizu MH, Berretta A, Teles F, Noronha IL, Andrade L. Green propolis extract attenuates acute kidney injury and lung injury in a rat model of sepsis. Sci Rep. 2021 Mar 15;11(1):5925. doi: 10.1038/s41598-021-85124-6. PMID 33723330
- [Background] Silveira MAD, Teles F, Berretta AA, Sanches TR, Rodrigues CE, Seguro AC, Andrade L. Effects of Brazilian green propolis on proteinuria and renal function in patients with chronic kidney disease: a randomized, double-blind, placebo-controlled trial. BMC Nephrol. 2019 Apr 25;20(1):140. doi: 10.1186/s12882-019-1337-7. PMID 31023272
- [Background] Silveira MAD, De Jong D, Berretta AA, Galvao EBDS, Ribeiro JC, Cerqueira-Silva T, Amorim TC, Conceicao LFMRD, Gomes MMD, Teixeira MB, Souza SP, Santos MHCAD, San Martin RLA, Silva MO, Lirio M, Moreno L, Sampaio JCM, Mendonca R, Ultchak SS, Amorim FS, Ramos JGR, Batista PBP, Guarda SNFD, Mendes AVA, Passos RDH; BeeCovid Team. Efficacy of Brazilian green propolis (EPP-AF(R)) as an adjunct treatment for hospitalized COVID-19 patients: A randomized, controlled clinical trial. Biomed Pharmacother. 2021 Jun;138:111526. doi: 10.1016/j.biopha.2021.111526. Epub 2021 Mar 20. PMID 34311528
- [Background] Berretta AA, Silveira MAD, Condor Capcha JM, De Jong D. Propolis and its potential against SARS-CoV-2 infection mechanisms and COVID-19 disease: Running title: Propolis against SARS-CoV-2 infection and COVID-19. Biomed Pharmacother. 2020 Nov;131:110622. doi: 10.1016/j.biopha.2020.110622. Epub 2020 Aug 17. PMID 32890967
- [Background] Maruta H, He H. PAK1-blockers: Potential Therapeutics against COVID-19. Med Drug Discov. 2020 Jun;6:100039. doi: 10.1016/j.medidd.2020.100039. Epub 2020 Apr 19. PMID 32313880
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Machado JL, Assuncao AK, da Silva MC, Dos Reis AS, Costa GC, Arruda Dde S, Rocha BA, Vaz MM, Paes AM, Guerra RN, Berretta AA, do Nascimento FR. Brazilian green propolis: anti-inflammatory property by an immunomodulatory activity. Evid Based Complement Alternat Med. 2012;2012:157652. doi: 10.1155/2012/157652. Epub 2012 Dec 19. PMID 23320022
- [Background] Shimizu T, Hino A, Tsutsumi A, Park YK, Watanabe W, Kurokawa M. Anti-influenza virus activity of propolis in vitro and its efficacy against influenza infection in mice. Antivir Chem Chemother. 2008;19(1):7-13. doi: 10.1177/095632020801900102. PMID 18610553
- [Background] Ito J, Chang FR, Wang HK, Park YK, Ikegaki M, Kilgore N, Lee KH. Anti-AIDS agents. 48.(1) Anti-HIV activity of moronic acid derivatives and the new melliferone-related triterpenoid isolated from Brazilian propolis. J Nat Prod. 2001 Oct;64(10):1278-81. doi: 10.1021/np010211x. PMID 11678650
- [Background] Berretta AA, Nascimento AP, Bueno PC, Vaz MM, Marchetti JM. Propolis standardized extract (EPP-AF(R)), an innovative chemically and biologically reproducible pharmaceutical compound for treating wounds. Int J Biol Sci. 2012;8(4):512-21. doi: 10.7150/ijbs.3641. Epub 2012 Mar 21. PMID 22457606
- [Derived] Silveira MAD, Menezes MA, de Souza SP, Galvao EBDS, Berretta AA, Caldas J, Teixeira MB, Gomes MMD, Damiani LP, Bahiense BA, Cabral JB, De Oliveira CWLM, Mascarenhas TR, Pinheiro PCG, Alves MS, de Melo RMV, Leite FM, Nonaka CKV, Souza BSF, Baptista NU, Teles F, da Guarda SF, Mendes AVA, Passos RDH. Standardized Brazilian green propolis extract (EPP-AF(R)) in COVID-19 outcomes: a randomized double-blind placebo-controlled trial. Sci Rep. 2023 Oct 27;13(1):18405. doi: 10.1038/s41598-023-43764-w. PMID 37891178
- [Derived] Silveira MAD, de Souza SP, Dos Santos Galvao EB, Teixeira MB, Gomes MMD, Damiani LP, Bahiense BA, Cabral JB, De Oliveira CWLM, Mascarenhas TR, Pinheiro PCG, Alves MS, de Melo RMV, Berretta AA, Leite FM, Nonaka CKV, de Freitas Souza BS, Mendes AVA, da Guarda SF, da Hora Passos R. The use of standardized Brazilian green propolis extract (EPP-AF) as an adjunct treatment for hospitalized COVID-19 patients (BeeCovid2): a structured summary of a study protocol for a randomized controlled trial. Trials. 2022 Apr 4;23(1):255. doi: 10.1186/s13063-022-06176-1. PMID 35379306